CLINICAL TRIAL: NCT02488434
Title: The Effectiveness of Using Fertile Chip on Intracytoplasmic Sperm Injection Undergoing Ivf Programme in Unexplained Infertile Couples
Brief Title: The Effects of Using Fertile Chip in Sperm Selection for Intracytoplasmic Sperm Injection in Unexplained Infertility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Selçuk Yetkinel, Clinical Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA15/132
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Unexplained Infertility
Keywords: ICSI; sperm selection; fertile chip; ıcsı outcomes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fertile chip (Active Comparator): sperm selection by using fertile chip and conventional methods
  Interventions: Device: fertile chip
- classical ICSI procedure (No Intervention): unexplained infertile couples who will be undertaken intracytoplasmic sperm injection (ICSI) for fertilisation

INTERVENTIONS:
Device: fertile chip — a new method for sperm selection on ivf cycles by using microchannel system.
  Arms: fertile chip

SUMMARY:
The aim of the current study is to evaluate to effectiveness of sperm selection by using fertile chip in unexplained infertile couples on intracytoplasmic sperm injection (ICSI) cycles.

DETAILED DESCRIPTION:
The aim of the current study is to evaluate to effectiveness of sperm selection by using fertile chip in unexplained infertile couples on intracytoplasmic sperm injection (ICSI) cycles. On study arm sperm selection will be performed by using special microchannel system which is called fertile chip (FC) without using sperm wash procedure. This FC system leads to select lineer motile progressive sperm selection. In control group, sperm selection will be performed by classical way which sperm will be undertaken to sperm wash by gradient method.

After selection of sperm in both arms, ICSI will be performed. The outcomes of ICSI schedule will be assesed by fertilization and clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* between 20-37 year-old women
* normal tubal patency, normal uterine cavity, normal ovulation,
* between 20-40 year-old men
* normal semen analyse by WHO criterias
* unexplained infertile couples

Exclusion Criteria:

* poor ovarian reserve which is diagnosed by Bologna criterias
* abnormal semen analyse by WHO sperm criterias
* abnormal ovulation problems,tubal patency or uterine cavity

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
increase fertilisation rate | 2 days

SECONDARY OUTCOMES:
Clinical pregnancy rates | 10 months

OTHER OUTCOMES:
The number of freezing embryos | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Esra Bulgan Kılıçdağ, MD, Study Director — Division of Reproductive and Endocrinology Unit, Department of Obstetrics and Gynecology, Faculty of Medicine, Baskent University, Adana, Turkey
Locations (1):
- Baskent University Faculty of Medicine Department of Obstetrics and Gynecology Division of Reproductive and Endocrinology Unit, Adana, Yüreğir, Turkey (Türkiye)

REFERENCES:
- [Background] Collins JA, Crosignani PG. Unexplained infertility: a review of diagnosis, prognosis, treatment efficacy and management. Int J Gynaecol Obstet. 1992 Dec;39(4):267-75. doi: 10.1016/0020-7292(92)90257-j. PMID 1361459
- [Background] Templeton AA, Penney GC. The incidence, characteristics, and prognosis of patients whose infertility is unexplained. Fertil Steril. 1982 Feb;37(2):175-82. doi: 10.1016/s0015-0282(16)46035-8. PMID 7060767
- [Background] Zini A, Finelli A, Phang D, Jarvi K. Influence of semen processing technique on human sperm DNA integrity. Urology. 2000 Dec 20;56(6):1081-4. doi: 10.1016/s0090-4295(00)00770-6. PMID 11113773
- [Background] Asghar W, Velasco V, Kingsley JL, Shoukat MS, Shafiee H, Anchan RM, Mutter GL, Tuzel E, Demirci U. Selection of functional human sperm with higher DNA integrity and fewer reactive oxygen species. Adv Healthc Mater. 2014 Oct;3(10):1671-9. doi: 10.1002/adhm.201400058. Epub 2014 Apr 17. PMID 24753434
- [Background] Moghissi KS, Wallach EE. Unexplained infertility. Fertil Steril. 1983 Jan;39(1):5-21. doi: 10.1016/s0015-0282(16)46750-6. PMID 6336697
- [Background] Practice Committee of the American Society for Reproductive Medicine. Definitions of infertility and recurrent pregnancy loss. Fertil Steril. 2008 Jun;89(6):1603. doi: 10.1016/j.fertnstert.2008.03.002. Epub 2008 May 16. No abstract available. PMID 18485348
- [Derived] Yetkinel S, Kilicdag EB, Aytac PC, Haydardedeoglu B, Simsek E, Cok T. Effects of the microfluidic chip technique in sperm selection for intracytoplasmic sperm injection for unexplained infertility: a prospective, randomized controlled trial. J Assist Reprod Genet. 2019 Mar;36(3):403-409. doi: 10.1007/s10815-018-1375-2. Epub 2018 Dec 12. PMID 30542782
- See also: fertile chip official site — http://fertilechip.com/en/